CLINICAL TRIAL: NCT07003399
Title: Diaphragmatic Morphofunction and Respiratory Drive in OSA and COPD: Insights From Ultrasound and EMG-based Cross-Sectional Analysis
Brief Title: Diaphragmatic Function and Respiratory Drive in OSA and COPD
Status: Recruiting | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Ning Ding, Principal Investigator, Nanjing Medical University
Other Study IDs: 2021-SR-347
Record Dates: First submitted 2025-05-15; First posted 2025-06-04 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Chronic Obstructive Pulmonary Disease; Overlap Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Normal Group: Healthy subjects with no known respiratory diseases or sleep disorders, serving as the control group for baseline comparison of diaphragmatic function and respiratory drive.
  Interventions: Other: Diaphragmatic Ultrasound and EMG Assessment
- OSA Group: Patients diagnosed with obstructive sleep apnea (OSA) based on polysomnography criteria (AHI ≥ 5 events/hour), evaluated for diaphragmatic function and respiratory drive using ultrasound and EMG.
  Interventions: Other: Diaphragmatic Ultrasound and EMG Assessment
- COPD Group: Patients diagnosed with chronic obstructive pulmonary disease (COPD) based on GOLD guidelines, assessed for diaphragmatic morphofunction and respiratory drive.
  Interventions: Other: Diaphragmatic Ultrasound and EMG Assessment
- Overlap Group: Patients with overlap syndrome (coexisting OSA and COPD), evaluated for diaphragmatic function and respiratory drive using ultrasound and EMG to explore combined disease impact.
  Interventions: Other: Diaphragmatic Ultrasound and EMG Assessment

INTERVENTIONS:
Other: Diaphragmatic Ultrasound and EMG Assessment — Non-invasive assessment of diaphragmatic morphofunction and respiratory drive using ultrasound imaging and diaphragm electromyography (EMG). This evaluation will be performed once per participant without any therapeutic intervention.

SUMMARY:
This cross-sectional observational study aims to assess the diaphragmatic morphofunction and respiratory drive characteristics among patients with obstructive sleep apnea (OSA), chronic obstructive pulmonary disease (COPD), overlap syndrome (OS), and healthy controls. Using ultrasound imaging and surface diaphragm electromyography (EMGdi), the study will explore group differences in diaphragmatic morphology, function, and respiratory drive indicators, and evaluate their clinical significance in disease differentiation and severity assessment.

DETAILED DESCRIPTION:
This is a single-center cross-sectional study designed to compare the diaphragmatic morphofunction and respiratory drive among four groups: OSA, COPD, overlap syndrome (patients with both OSA and COPD), and healthy controls. Participants will undergo overnight polysomnography (PSG), spirometry, impulse oscillometry, and diaphragm ultrasound combined with surface EMGdi measurements. The study will analyze group differences in diaphragmatic thickness, excursion, thickening fraction, and EMGdi parameters including EMGdi-rest, EMGdi-max, and EMGdi%max. The relationships between diaphragmatic indicators and respiratory parameters (FEV1, FVC, AHI, R5-R20, etc.) will also be assessed. This study aims to provide objective evidence for diaphragmatic dysfunction characterization in OSA and COPD, as well as to explore its diagnostic utility in overlap syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 18 and 80 years.
2. For OSA Group: Diagnosed obstructive sleep apnea with AHI ≥ 5 events/hour based on overnight polysomnography.
3. For COPD Group: Diagnosed chronic obstructive pulmonary disease based on GOLD guidelines.
4. For Overlap Group: Diagnosed both OSA (AHI ≥ 5) and COPD.
5. For Control Group: Healthy volunteers with no known respiratory diseases or sleep disorders.
6. Ability and willingness to provide informed consent for participation in the study.

Exclusion Criteria:

1. Severe cardiovascular diseases (e.g., unstable angina, heart failure NYHA III/IV).
2. Severe hepatic or renal insufficiency.
3. Neuromuscular diseases affecting respiratory muscles.
4. Recent upper airway or thoracic surgery (within 3 months).
5. Pregnancy or breastfeeding.
6. Participants who cannot complete assessments due to cognitive impairment or poor cooperation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with obstructive sleep apnea, chronic obstructive pulmonary disease, overlap syndrome (OSA and COPD), and healthy volunteers from a single center. Subjects will be evaluated for diaphragmatic morphofunction and respiratory drive using ultrasound and EMG.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Diaphragmatic electromyography (EMGdi-rest) at baseline | Baseline (at enrollment)
  To assess resting diaphragmatic electromyographic activity (µV) across OSA, COPD, Overlap, and control groups using surface and esophageal EMG.
Diaphragmatic EMG during maximal inspiration (EMGdi-max) | Baseline (at enrollment)
  To assess maximal inspiratory diaphragmatic EMG activity (µV) using voluntary effort tests with surface and esophageal EMG.
Relative inspiratory EMG effort (EMGdi%max) | Baseline (at enrollment)
  To calculate the ratio of EMGdi-rest to EMGdi-max as a percentage, reflecting the relative inspiratory effort.

SECONDARY OUTCOMES:
Diaphragmatic excursion measured by ultrasound during deep breathing | Baseline (at enrollment)
  To evaluate diaphragmatic mobility (cm) during deep breathing using standardized ultrasound protocols.
Respiratory impedance parameter R5 | Baseline (at enrollment)
  To compare small airway resistance (kPa·s·L-¹) between groups using impulse oscillometry.
Respiratory resistance at 20 Hz (R20) | Baseline (at enrollment)
  To compare central airway resistance (kPa·s·L-¹) using impulse oscillometry.
Difference in resistance (R5-R20) | Baseline (at enrollment)
  To evaluate small airway dysfunction by calculating the difference between R5 and R20 (kPa·s·L-¹) .
Forced expiratory volume in 1 second (FEV1) | Baseline (at enrollment)
  To compare FEV1 (L) across groups and assess its relationship with diaphragmatic function.
Forced vital capacity (FVC) | Baseline (at enrollment)
  To compare FVC (L) across groups and assess pulmonary capacity.
FEV1/FVC ratio | Baseline (at enrollment)
  To evaluate airflow obstruction using the FEV1/FVC ratio (%).
Apnea-hypopnea index (AHI) | Baseline (at enrollment)
  To evaluate sleep-disordered breathing severity (events/hour) in OSA and Overlap groups.
Oxygen desaturation index (ODI) | Baseline (at enrollment)
  To assess oxygen desaturation frequency during sleep (events/hour) using PSG data.
Minimum oxygen saturation (SpO₂ min) | Baseline (at enrollment)
  To capture the lowest oxygen saturation (%) during overnight monitoring.
Time below 90% oxygen saturation (T90) | Baseline (at enrollment)
  To calculate the percentage of sleep time with oxygen saturation < 90% (%).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared. The informed consent will be ansigned before enrolled in the study and ensured to keep personal information confidential.

REFERENCES:
- [Background] Domnik NJ, Phillips DB, James MD, Ayoo GA, Taylor SM, Scheeren RE, Di Luch AT, Milne KM, Vincent SG, Elbehairy AF, Crinion SJ, Driver HS, Neder JA, O'Donnell DE. Compensatory responses to increased mechanical abnormalities in COPD during sleep. Eur J Appl Physiol. 2022 Mar;122(3):663-676. doi: 10.1007/s00421-021-04869-0. Epub 2022 Jan 16. PMID 35034195
- [Background] Jolley C, Luo Y, Steier J, Sylvester K, Man W, Rafferty G, Polkey M, Moxham J. Neural respiratory drive and symptoms that limit exercise in chronic obstructive pulmonary disease. Lancet. 2015 Feb 26;385 Suppl 1:S51. doi: 10.1016/S0140-6736(15)60366-X. PMID 26312873
- [Background] He BT, Lu G, Xiao SC, Chen R, Steier J, Moxham J, Polkey MI, Luo YM. Coexistence of OSA may compensate for sleep related reduction in neural respiratory drive in patients with COPD. Thorax. 2017 Mar;72(3):256-262. doi: 10.1136/thoraxjnl-2016-208467. Epub 2016 Nov 2. PMID 27807016
- [Background] Zhang N, Luo Y, Yang L, Liu Z, Qiu Z, Huang Q, Zhang Y. Novel method for evaluating the upper airway resistance using the ratio of neural respiratory drive to flow in OSA. Sleep Med. 2020 Sep;73:162-169. doi: 10.1016/j.sleep.2020.05.006. Epub 2020 May 15. PMID 32836084
- [Background] Ramsook AH, Koo R, Molgat-Seon Y, Dominelli PB, Syed N, Ryerson CJ, Sheel AW, Guenette JA. Diaphragm Recruitment Increases during a Bout of Targeted Inspiratory Muscle Training. Med Sci Sports Exerc. 2016 Jun;48(6):1179-86. doi: 10.1249/MSS.0000000000000881. PMID 26795460
- [Background] James MD, Phillips DB, Vincent SG, Abdallah SJ, Donovan AA, de-Torres JP, Neder JA, Smith BM, Jensen D, O'Donnell DE; Canadian Respiratory Research Network. Exertional dyspnoea in patients with mild-to-severe chronic obstructive pulmonary disease: neuromechanical mechanisms. J Physiol. 2022 Sep;600(18):4227-4245. doi: 10.1113/JP283252. Epub 2022 Aug 5. PMID 35861594